CLINICAL TRIAL: NCT05195229
Title: Quantifying Viral Load in Respiratory Particles That Are Generated by Children and Adults With COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas B. Kinane, M.D, MD Pediatric Medical Services (MGHfC), Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020P002886
Record Dates: First submitted 2022-01-13; First posted 2022-01-18 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19; Viral Load
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Aim: To estimate the viral load in aerosols generated from children with COVID-19 infection, and to compare the viral load contained in aerosols from children with aerosols from adults
  Interventions: Device: COVID-19 Aerosol Collection

INTERVENTIONS:
Device: COVID-19 Aerosol Collection — Step 1: A nasal and oral swab will be obtained to establish the nasopharyngeal viral load.
  Step 2: Study staff will use the CCI and/or UPAS to collect aerosol samples for viral load. Staff will sample the room aerosol for 30 minutes while the participant does not wear a mask, and then if the participant is interested, staff will sample room aerosol while the participant wears different types of masks. If the participant does not tolerate wearing a surgical mask, or if the providers believe this is contraindicated, researchers will forego this portion of the study procedures. If an accompanying family member chooses to stay in the patient room during testing, they will be provided with an N95 respirator.

SUMMARY:
The study will be a prospective cohort design to determine if children generate aerosols that harbor a viral load similar to adults. Prior to beginning enrollment, researchers may recruit up to 10 participants (adults or children who meet inclusion criteria for the main study) to perform a small pilot to optimize our cold chain and laboratory procedures.

The study will include children and adults who are confirmed SARS-CoV-2 positive and aim for a total sample size of at least 10 children and 10 adults.

Hypothesis: As children have a high viral load in the nasopharynx, we hypothesize that children generate aerosols that contain SARS-CoV-2 virus.

Aim: To estimate the viral load in aerosols generated from children with COVID-19 infection, and to compare the viral load contained in aerosols from children with aerosols from adults

DETAILED DESCRIPTION:
For children and adults who are admitted to MGH, study staff will perform:

Step 1: A nasal and oral swab will be obtained to establish the nasopharyngeal viral load.

Step 2: Study staff will use the CCI and/or UPAS to collect aerosol samples for viral load. Staff will sample the room aerosol for 30 minutes while the participant does not wear a mask, and then if the participant is interested, staff will sample room aerosol while the participant wears different types of masks. If the participant does not tolerate wearing a surgical mask, or if the providers believe this is contraindicated, researchers will forego this portion of the study procedures. If an accompanying family member chooses to stay in the patient room during testing, they will be provided with an N95 respirator.

Step 3: Staff will ask participants to repeat these steps and provide a sample each day that they are having symptoms of COVID-19. The study may conduct serial sampling, where participants could be asked to provide a sample each day that they are having symptoms of COVID-19 up until discharge, or once symptoms resolve. Once symptoms resolve or the patient is discharged, sampling will be complete.

ELIGIBILITY:
Inclusion criteria:

* SARS-CoV-2 PCR positive in the last fourteen days
* Symptomatic with typical symptoms of COVID-19, including fever, cough, nasal congestion, rhinorrhea, anosmia, ageusia, shortness of breath, chest pain, fatigue, myalgias, or other atypical symptoms with documentation of that symptom OR
* Asymptomatic with laboratory confirmation of cycle threshold value < 30.

Exclusion criteria:

* Chronic respiratory disease or neuromuscular condition associated with severely reduced lung function defined as FEV1 or FVC <50% predicted, or requiring chronic supplemental oxygen or respiratory support
* On current respiratory support via supplemental oxygen, non-invasive ventilation, or invasive mechanical ventilation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Viral Load in Aerosols generated from COVID-19 | 10 days
  The viral load in aerosols generated from children with COVID-19 infection, and to compare the viral load contained in aerosols from children with aerosols from adults. Measures will be extracted to assess if the cycle threshold value is high enough in aerosols for virus to be transmitted to others.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Kinane, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No